CLINICAL TRIAL: NCT01330732
Title: The Correlation Between Radiological Evaluation of Kyphosis and Evaluation Using SPINESCAN®
Brief Title: Kyphosis Evaluation Using SPINESCAN®
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Yoram Anekstein, MD, Assaf-Harofeh Medical Center
Other Study IDs: 109/08
Record Dates: First submitted 2009-03-15; First posted 2011-04-07 (Estimated); Last update posted 2011-04-07 (Estimated); Status verified 2008-08

CONDITIONS: Kyphosis
Keywords: SPINESCAN®; kyphosis
MeSH Terms: conditions — Kyphosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Main group: patients examined in scoliosis clinic for kyphosis with recent lateral spine X-rays.

SUMMARY:
The purpose of this study is to evaluate the accuracy of SPINESCAN® with standard lateral x-rays of the spine in patients monitored for kyphosis.

DETAILED DESCRIPTION:
Kyphosis is usually a developmental deformity of the spine in the sagittal plane. Once diagnosed, serial X-rays are used for followup. These are usually required at yearly intervals.

SPINESCAN® is a computerized digital inclinometer, design for evaluating angular spine deformities.

Patients examined in the spine clinic with recent X-rays will be examined with SPINESCAN® and it's results compared with the classical radiological assessment.

ELIGIBILITY:
Inclusion Criteria:

* Patients examined in scoliosis clinic for kyphosis with recent lateral spine X-rays.
* Age: 7 years old and above.

Exclusion Criteria:

* Less than 7 years old.
* No informed consent.

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Main group: patients examined in scoliosis clinic for kyphosis with recent lateral spine X-rays.
  Age: 7 and above.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-11 (Estimated); Study Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
Kyphosis degree (by SPINESCAN®) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yigal Mirovsky, MD, Study Chair — Assaf-Harofeh Medical Center
Locations (1):
- Assaf HaRofeh Medical Center, Ẕerifin, Israel

REFERENCES:
- [Background] Ovadia D, Bar-On E, Fragniere B, Rigo M, Dickman D, Leitner J, Wientroub S, Dubousset J. Radiation-free quantitative assessment of scoliosis: a multi center prospective study. Eur Spine J. 2007 Jan;16(1):97-105. doi: 10.1007/s00586-006-0118-8. Epub 2006 May 17. PMID 16705434